CLINICAL TRIAL: NCT02685189
Title: Long-Term Clinical Follow-Up of Children Enrolled in Stannsoporfin Clinical Trial Protocol No. 64,185-06-2(W)(WS)(ISNHP)
Brief Title: Long-Term Clinical Follow-Up of Children Enrolled in Stannsoporfin Clinical Trial Protocol No. 64,185-06-2(W)
Status: Terminated | Type: Observational
Why Stopped: Study stopped for business reasons and not for any safety reasons.
Sponsor: InfaCare Pharmaceuticals Corporation, a Mallinckrodt Company (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Other Study IDs: 64,185-06LT-2
Record Dates: First submitted 2016-02-10; First posted 2016-02-18 (Estimated); Last update posted 2019-10-15 (Actual); Status verified 2016-02

CONDITIONS: Hyperbilirubinemia
MeSH Terms: conditions — Hyperbilirubinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 0.75 mg/kg Previous exposure to stannsoporfin: Previous exposure 0.75 mg/kg
  Interventions: Other: Previous exposure to stannsoporfin
- 1.5 mg/kg Previous exposure to stannsoporfin: Previous exposure 1.5 mg/kg
  Interventions: Other: Previous exposure to stannsoporfin

INTERVENTIONS:
Other: Previous exposure to stannsoporfin — No intervention in this protocol

SUMMARY:
The purpose of this protocol is to provide a mechanism to collect Long Term Clinical Data from those babies who participated in the primary Study 64,185-06-2(W)(WS)(ISNHP) "An Open-Label Study Of The Safety And Clinical Pharmacology Of Stanate® In Infants At-Risk For Exchange Transfusion".

DETAILED DESCRIPTION:
The purpose of this protocol is to provide a mechanism to collect Clinical Data from those babies who participated in the primary Study 64,185-06-2(W)(WS)(ISNHP) "An Open-Label Study Of The Safety And Clinical Pharmacology Of Stanate® In Infants At-Risk For Exchange Transfusion". Data on long-term impact of Stannsoporfin on the physical, neurological, neurodevelopmental, biochemical, metabolic and hematopoietic profiles of the children will be collected at 9 and 18 months, 3, 6 and 9 years after Stannsoporfin administration

ELIGIBILITY:
Inclusion Criteria:

* All children who have been enrolled and received Stanate® Injection/Placebo in Study Protocol 64,185-06-2(W)(WS)(ISNHP) are eligible for this follow-up.

Exclusion Criteria:

-

Ages: 1 Day to 60 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All children who have been enrolled and received Stanate® Injection/Placebo in Study Protocol 64,185-06-2(W)(WS)(ISNHP) are eligible for this follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2006-07; Primary Completion 2016-05-10 (Actual); Study Completion 2016-05-10 (Actual)

PRIMARY OUTCOMES:
NEUROLOGICAL EXAMINATION; Child Behavior Check List | 10 years
  Child Behavior Check List is a standardized measure in child psychology for evaluating maladaptive behavioral and emotional problems in preschool patients

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Ruiz, MD, Study Director — InfaCare Pharmaceuticals Corporation, a Mallinckrodt Company